CLINICAL TRIAL: NCT00365547
Title: Phase II Clinical Study of Weekly Topotecan in Combination With Avastin™ in Patients With Stage IIIB/IV Non-Small Cell Lung Cancer Who Have Failed Prior Systemic Chemotherapy
Brief Title: Topotecan and Bevacizumab in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer That Did Not Respond to Previous Systemic Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005LS083; UMN-0602M81427 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2012-06-15 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Bevacizumab; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients Treated With Topotecan and Avastin in NSCLC (Experimental): Weekly topotecan hydrochloride and bi-weekly Avastin (bevacizumab) in patients with non-small cell lung cancer (NSCLC) who have failed prior systemic chemotherapy.
  Interventions: Biological: bevacizumab; Drug: topotecan hydrochloride

INTERVENTIONS:
Biological: bevacizumab — Will be given by intravenous (IV) infusion at the dose of 10 mg/kg on days 1 and 15 after topotecan administration until disease progression or for another reason.
  Other Names: Avastin
Drug: topotecan hydrochloride — Topotecan 4 mg/m^2 intravenously (IV) will be given as a 30-minute intravenous infusion on days 1, 8, and 15 with a rest on day 22. Treatment will be repeated every 28 days until disease progression or for another reason.
  Other Names: Hycamtin(TM)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as Avastin (bevacizumab), can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving topotecan together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving topotecan together with bevacizumab works in treating patients with stage IIIB or stage IV non-small cell lung cancer that did not respond to previous systemic chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the progression-free survival of patients with stage IIIB or IV non-small cell lung cancer treated with topotecan hydrochloride and bevacizumab who have failed prior systemic chemotherapy.

Secondary

* Determine the objective response rates in patients treated with this regimen.
* Measure time-to-event efficacy variables, including time to objective tumor response (for responding patients), duration of response (for responding patients), time to treatment failure, and overall survival.
* Characterize the quantitative and qualitative toxicities of this regimen in these patients.

OUTLINE: Patients receive topotecan hydrochloride intravenously (IV) over 30 minutes on days 1, 8, and 15 and Avastin (bevacizumab) IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 6 months from registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-small cell lung cancer (NSCLC). Patients with extrathoracic-only squamous cell NSCLC are eligible. Intrathoracic squamous cell carcinoma will not be eligible. Mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible.
* Disease that has failed one or more prior standard therapy and is no longer likely to respond to such therapy.
* Prior systemic chemotherapy, immunotherapy, or biological therapy is allowed, except for prior use of Avastin and topotecan in combination. Patient must be at least 14 days from previous radiation or systemic therapy (at least 30 days for investigational agents) and have recovered from the acute toxic effects of the treatment prior to study enrollment.
* Disease status must be measurable or evaluable as defined by Response Evaluation Criteria In Solid Tumors (RECIST criteria)
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1
* Age 18 years or greater
* Adequate organ function within 14 days of study registration including the following:

  * Adequate bone marrow reserve:

    * absolute neutrophil count (ANC) > or = to 1.5 x 10^9/L,
    * platelets >100 x 10^9/L,
    * hemoglobin > 9 g/dL
  * Hepatic:

    * bilirubin <1.5 times the upper limit of normal (x ULN),
    * alkaline phosphatase (ALP), aspartate transaminase (AST) and alanine transaminase (ALT) <3.0 x ULN (ALP, AST, and ALT <5 x ULN is acceptable if liver has tumor involvement)
  * Renal:

    * serum creatinine < 2.0
    * urine dipstick for proteinuria < 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible)
  * Coagulation:

    * International Normalized Ratio (INR) < 1.5
    * Partial thromboplastin time (PTT) < the upper limits of normal (ULN)
* Women of childbearing potential and sexually active males are required to use an effective method of contraception (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the study and for 3 months after the last dose of study drug.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Pregnant (positive pregnancy test) or breast-feeding. Topotecan is pregnancy category D - clear evidence of risk in pregnancy; Avastin is pregnancy category C - risk in pregnancy cannot be ruled out. Pregnancy testing is not required for post-menopausal or surgically sterilized women
* Known hypersensitivity to any component of Avastin (bevacizumab)
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Known central nervous system (CNS) disease, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (≥ ½ teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Active malignancy other than non-small cell lung cancer (NSCLC), treated superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within last five years are allowed.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Dudek, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 patients were enrolled, only 43 patients received study medication
Groups:
- Intent-To-Treat Population: Patients who enrolled and were scheduled to receive weekly topotecan (4 mg/m^2 will be given as a 30-minute intravenous infusion on days 1, 8, and 15 with a rest on day 22 and repeated every 28 days) and bi-weekly Avastin (bevacizumab given by IV infusion at the dose of 10 mg/kg on days 1 and 15 after topotecan administration)in patients with non-small cell lung cancer (NSCLC) who have failed prior systemic chemotherapy.
Period: Overall Study
Arm/Group | Intent-To-Treat Population
Started | 46
Completed | 43
Not Completed | 3
Not completed — Insurance did not cover Avastin | 1
Not completed — Screen failure | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intent-To-Treat Population
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Disease Progression
Description: Assessed by Response Evaluation Criteria In Solid Tumor (RECIST criteria). Progression is defined as a measureable increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions since baseline.
Time Frame: From Day 1 Until First Documented Disease Progression or Date of Death (Whichever Occurred First)
Population: All intent-to-treat patients enrolled were analyzed. Maximum number of days was 1349.
Measure: Mean (95% Confidence Interval); unit: Days
Groups:
- Intent-To-Treat Population: Patients who enrolled and were scheduled to receive weekly topotecan (4 mg/m^2 will be given as a 30-minute intravenous infusion on days 1, 8, and 15 with a rest on day 22 and repeated every 28 days) and bi-weekly Avastin (bevacizumab) given by intravenous (IV) infusion at the dose of 10 mg/kg on days 1 and 15 after topotecan administration)in patients with non-small cell lung cancer (NSCLC) who have failed prior systemic chemotherapy.
Arm/Group | Intent-To-Treat Population
Number analyzed (Participants) | 46
Days | 152 [112 to 233]

2. Secondary Outcome: Number of Tumor Responders
Description: Patients that met Solid Tumor Response Criteria (RECIST) criteria for partial response (at least a 30% decrease in the sum of the longest diameters of target lesions) and complete response (disappearance of all target lesions).
Time Frame: From Day 1 Until Disease Progression or Date of Death (Whichever Occurred First), Up to 1 Year
Measure: Number; unit: Participants
Groups:
- Patients Evaluable for Tumor Response: Only patients that remained in the study for at least 2 months and had the tumor measurements necessary to meet RECIST criteria are included.
Arm/Group | Patients Evaluable for Tumor Response
Number analyzed (Participants) | 41
Participants
  Partial Response | 6
  Complete Response | 0

3. Secondary Outcome: Median Time to Response
Description: Defined as the time from the start of treatment until first documented evidence of at least a partial tumor response.
Time Frame: From Day 1 Until Tumor Response
Population: Maximum number of days for analysis was 104.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Patients Evaluable for Tumor Response: Patients that met Solid Tumor Response Criteria (RECIST) criteria for partial response (at least a 30% decrease in the sum of the longest diameters of target lesions) and complete response (disappearance of all target lesions).
Arm/Group | Patients Evaluable for Tumor Response
Number analyzed (Participants) | 6
Days | 62.5 [55 to 104]

4. Secondary Outcome: Median Duration of Response
Description: Defined to be the time from first documented evidence of response until the first documented sign of disease progression or death due to progressive disease. For subjects who do not progress or die, duration of response will be censored at the time of last contact.
Time Frame: Day of 1st Response Until Disease Progression of Death/Last Contact
Population: Maximum number of days was 1277.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Patients Evaluable for Tumor Response
Number analyzed (Participants) | 6
Days | 186.5 [105 to 1277]

5. Secondary Outcome: Median Overall Survival
Description: Defined as the time from the start of treatment until death due to whatever cause. For subjects alive at study completion, time to death will be censored at the time of last contact.
Time Frame: From Day 1 Until Death Occurred
Population: Maximum number of days was 1349.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Intent-To-Treat Population
Number analyzed (Participants) | 46
Days | 345 [213 to 464]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from Day 1 of treatment through 4 weeks post treatment. AEs were not collected for 3 patients who were enrolled but never received treatment.
Groups:
- Safety Population: Patients who received treatment with weekly topotecan (4 mg/m^2 will be given as a 30-minute intravenous infusion on days 1, 8, and 15 with a rest on day 22 and repeated every 28 days) and bi-weekly Avastin (bevacizumab given by IV infusion at the dose of 10 mg/kg on days 1 and 15 after topotecan administration)in patients with non-small cell lung cancer (NSCLC) who have failed prior systemic chemotherapy.
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 10/43
Other Adverse Events (participants affected / at risk) | 36/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=43)
Pain, muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Infection with normal ANC or G1/2 neutrophils-blood (Infections and infestations) | 1 (1)
Infection with normal ANC or G1/2 neutrophils - lung (Infections and infestations) | 1 (1)
Fever in absence of neutropenia (General disorders) | 1 (1)
Progressive disease (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage, pulmonary (Blood and lymphatic system disorders) | 1 (1)
Pain, pleura (General disorders) | 1 (1)
Pain, abdomen (General disorders) | 1 (1)
Obstruction, small bowel (Gastrointestinal disorders) | 1 (1)
Pain, chest wall (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pain, bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=43)
Achy, muscle aches (Musculoskeletal and connective tissue disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 11 (25)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Fatigue (General disorders) | 17 (28)
Headache (General disorders) | 12 (13)
Upper respiratory infection (Infections and infestations) | 3 (4)
Malaise (General disorders) | 3 (12)
Neutropenia (Blood and lymphatic system disorders) | 6 (8)
Nausea (Gastrointestinal disorders) | 17 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Rib pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Chest pain (General disorders) | 3 (3)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Congestion, sinus/nasal (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (31)
Vomiting (Gastrointestinal disorders) | 5 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (18)
Epitaxis (Gastrointestinal disorders) | 3 (5)
Dyspnea, shortness of breath (Respiratory, thoracic and mediastinal disorders) | 7 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes